CLINICAL TRIAL: NCT07405437
Title: General Dentists' Knowledge, Attitudes and Utilisation of Silver Diamine Fluoride for Caries Management in Children: A Multi-Region Survey
Brief Title: General Dentists' Knowledge, Attitudes and Clinical Usage of SDF
Acronym: GDPKAUSDF
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC25009
Record Dates: First submitted 2025-07-02; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Decay, Dental
Keywords: silver diamine fluoride; general dental practicioners; knowledge; attitude; utilisation
MeSH Terms: conditions — Dental Caries; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will look at how dentists in the UK are using Silver Diamine Fluoride (SDF) in their everyday practice. SDF is a liquid treatment that helps stop tooth decay. It's especially useful for treating children, as it can be applied quickly and without the need for drilling or needles. However, it seems that not many dentists are using SDF regularly, and this research aims to find out why.

The study will use an anonymous online survey to ask dentists about:

* How much they know about SDF and its benefits.
* Whether they use SDF in their practice and how they use it.
* What might stop them from using SDF, such as lack of training, cost, or concerns about how patients might feel about it.

The answers will be analysed to see what's working well and what's not when it comes to SDF use. The goal is to help dentists better understand and use this treatment, making it easier to manage tooth decay in children and improve their overall oral health.

ELIGIBILITY:
Inclusion Criteria:

* GDPs currently practicing in Lothian & Yorkshire
* General dental practitioners registered with the General Dental Council

Exclusion Criteria:

* General dental practioners out with Lothian and Yorkshire General dental practitioners who do not see paediatric patients.
* General dental practitioners who do not offer NHS services.
* General dental practitioners who are no longer practicing.
* Those on the specialist registers
* Other dental care professions or dental students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General dental practitioners in Lothian, Scotland and Yorkshire, England
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Awareness | Once only data collection day 1
  General dentists' awareness and perception survey
Knowledge | Once only data collection day 1
  General dentists' awareness and perception survey and applications of silver diamine fluoride
Utilisation | Once only data collection day 1
  General dentists' awareness and perception survey
Influencing factors | Once only data collection day 1
  General dentists' awareness and perception survey

SECONDARY OUTCOMES:
Compare the knowledge, attitude, and usage of SDF in Lothian & Yorkshire | Once only data collection day 1
  General dentists' awareness and perception survey

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom